CLINICAL TRIAL: NCT06956651
Title: 18-Month Clinical Evaluation of Self-Adhesive Flowable Giomer Compared to Conventional Flowable Giomer in Conservative Occlusal Restorations: A Randomized Clinical Trial
Brief Title: 18-Month Clinical Evaluation of Self-Adhesive Flowable Giomer Compared to Conventional Flowable Giomer in Conservative Occlusal Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Ayman Kamal, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13579
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Occlusal Caries
Keywords: self adhesive giomer; class I; clinical performance; Beautifil Flow; FIT SA; USPHS Criteria
MeSH Terms: interventions — Beautifil Flow Plus F00

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beautifil Flow Plus X F00 (Active Comparator): Conventional flowable giomer restorative material
  Interventions: Other: Beautifil Flow Plus F00
- FIT SA (Experimental): Self Adhesive Flowable giomer restoration
  Interventions: Other: FIT SA

INTERVENTIONS:
Other: FIT SA — Self Adhesive Flowable giomer restorative material
  Arms: FIT SA
Other: Beautifil Flow Plus F00 — Conventional Flowable giomer composite
  Arms: Beautifil Flow Plus X F00

SUMMARY:
The study compares two restorative materials to restore occlusal decay, offering the patients high-strength, high-durability restorations with antibacterial properties.

DETAILED DESCRIPTION:
There is no available evidence discussing the FIT SA restorative material in the restoration of occlusal lesions. This study aims to provide valuable insights into the clinical performance of this restorative material compared to the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Posterior vital tooth with Class I caries.

Exclusion Criteria:

* Teeth with clinical symptoms of pulpitis, such as spontaneous pain.
* Pain or sensitivity to pressure.
* Non-vital teeth.
* Fractured or cracked teeth.
* Endodontically treated teeth.
* Periodontally affected teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | 18 months
  Clinical performance using the Modified United States Public Health Service criteria, values: alpha (upper value - better outcome), charlie (lower value- worse outcome).

IPD SHARING:
Plan to Share IPD: Yes
There is no available evidence assessing FIT SA restorative material in occlusal cavity restoration. Therefore, the study aims to provide insights into its clinical performance regarding functional and aesthetic aspects.